CLINICAL TRIAL: NCT04299139
Title: Chiropractic Treatment of Arthrogenic Torticollis in Infants; a Retrospective Study on Outcome in 1000 Infants
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Schweinhardt Petra, PhD, Balgrist University Hospital
Other Study IDs: 2017-01022
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Arthrogenic Torticollis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: chiropractic treatment — There is no intervention. Data that has been collected during the time a patient was attending a chiropractor. This data will be evaluated

SUMMARY:
Patient data is collected from previously treated patients and entered into the Research Electronic Data Capture (REDCap).

DETAILED DESCRIPTION:
Already collected patient data (1995-2013) from a privat practice, is screened and entered into a individually design REDCap form.

ELIGIBILITY:
Inclusion Criteria:

* arthrogenic torticollis
* male or female age 3-12 month
* treatment was conducted between 01/1995-12/2013

Exclusion Criteria:

* uncompleted record
* decline of further use of patient data

Ages: 3 Months to 12 Months | Sex: All
Age Groups: Child
Study Population: Children between the age of 3-12 months
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Treatment outcome | 3-12 month of age
  Subjective treatment outcome after chiropractic care

CONTACTS AND LOCATIONS:
Overall Officials: Anke Langenfeld, PhD, Study Chair — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Not yet defined